CLINICAL TRIAL: NCT05004103
Title: The Efficacy of Cosmetic Products and Its Effects on Facial Skin Microbiome
Brief Title: Cosmetic Products and Facial Skin Microbiome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Collaborators: PT Paragon Technology and Innovation (Unknown)
Responsible Party: Principal Investigator, Prof. dr. Franciscus D. Suyatna, PhD, SpFK, Clinical Pharmacology Professor, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRSU.P.PTI/11/20/17.02
Record Dates: First submitted 2021-07-08; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Cosmetics Product Effects
Keywords: Skin Microbiome; Facial Skin Microbiome; MIcrobiome diversity

STUDY DESIGN:
Intervention Model Description: Pre-post study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin microbiome evaluation (Experimental): Female healthy volunteers applied cosmetic products (cleanser and moisturizer cream), the diversity of skin microbiome will be examined before and after using the products
  Interventions: Other: Cosmetic products application

INTERVENTIONS:
Other: Cosmetic products application — Female healthy volunteers applied cosmetic products (cleanser and moisturizer) in the morning and afternoon for 1 month. Seven days wash out period will be conducted prior study starts. The evaluation will be conducted before, two weeks after treatment starts, and at the end of the study.

SUMMARY:
The skin microbiome diversity in female healthy volunteers will be studied along with cosmetic products application in 1 month period. This study is also aimed to investigate the efficacy of cosmetic products on skin rejuvenation. .

DETAILED DESCRIPTION:
The study is conducted in COVID-19 pandemic era, thus every person involved in this study must follow health protocol for COVID-19.

The study procedure, consist of screening visit (D -7), 7-day wash out, baseline visit (D 0), first follow up ( D 14), and second follow up (D 28).

1. Screening visit: obtained Informed Consent, COVID-19 detection by swab RT-PCR, and inclusion and exclusion criteria, wash out product dispensing, and subject's diary dispensing.
2. Baseline visit: Investigator will check vital signs, facial skin value by Cutometer, Mexameter, Sebumeter, Corneometer, Colorimeter, Tewameter, dan pH meter, and kin taping by Corneofix tape. Investigational Products will dispensed in this visit for 2 weeks usage.
3. First follow up: Investigator will check vital signs and facial skin value. Investigational Products will dispensed in this visit for 2 weeks usage.
4. Second follow up: Investigator will check vital signs, facial skin value, and skin taping by Corneofix tape.

All adverse events (AEs) occurred during study will be recorded in Case Report Form.

ELIGIBILITY:
Inclusion Criteria:

1. female 18-35 years old
2. signed the informed consent

Exclusion Criteria:

1. infected by COVID-19
2. females with skin diseases on face and neck such as atopic dermatitis, skin allergy, acne with moderate and severe degree, seborrheic dermatitis, malignancy
3. females with ongoing skin treatments.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy females
Enrollment: 24 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-08-20 (Estimated)

PRIMARY OUTCOMES:
Microbiome diversity index | 28 days
  The amount and diversity of microbiota will be observed on facial skin before and after product application
Facial skin elasticity | 28 days
  The ratio between pliability/firmness and expressed in mm. The result before and after product application will be observed by cutometer.
Sebum unit of facial skin | 28 days
  Sebumeter unit (mcg/cm2) of facial skin before and after product application will be observed using sebumeter. This sebumeter unit reflects the concentration of sebum on skin per observed area.
Capacity of corneometer unit | 28 days
  Corneometer unit reflects the moist index of skin. The corneometer unit observed by Corneometer, before and after product application.
Skin color intensity | 28 dyas
  The skin color expressed in colorimeter index value. The observation is conducted before and after product application
Transepidermal Waterloss (g/h/m2) | 28 days
  The hydration of skin is observed by Tewameter. The observation is conducted before and after product application
pH of facial skin | 28 days
  The pH of facial skin is observed using skin-pH-meter. Observation is conducted before and after product application
The skin color related to the Minimal Erythema Dosage (MED) | 28 Days
  The skin color (MED) is observed using Mexameter and is conducted before and after product application

CONTACTS AND LOCATIONS:
Overall Officials: Frans Suyatna, Prof, PhD, Principal Investigator — Clinical Research Supporting Unit, Faculty of Medicine, University of Indonesia
Locations (1):
- Clinical Research Supporting Unit, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collins-Fulea C, Klima K, Wegienka GR. Prevalence of low vitamin D levels in an urban midwestern obstetric practice. J Midwifery Womens Health. 2012 Sep-Oct;57(5):439-44. doi: 10.1111/j.1542-2011.2012.00167.x. PMID 22954074
- [Background] Vijay A, Gupta S, Rawat S, Jain SK. A Rare Case of Coinfection with White Piedra and Pediculosis Capitis. Indian Dermatol Online J. 2017 Jul-Aug;8(4):279-280. doi: 10.4103/idoj.IDOJ_353_16. No abstract available. PMID 28761849
- [Background] Wallen-Russell, C. The Role of Every-Day Cosmetics in Altering the Skin Microbiome: A Study Using Biodiversity. Cosmetics 2019, 6, 2. https://doi.org/10.3390/cosmetics6010002
- [Result] Byrd AL, Belkaid Y, Segre JA. The human skin microbiome. Nat Rev Microbiol. 2018 Mar;16(3):143-155. doi: 10.1038/nrmicro.2017.157. Epub 2018 Jan 15. PMID 29332945
- [Result] Ogai K, Nagase S, Mukai K, Iuchi T, Mori Y, Matsue M, Sugitani K, Sugama J, Okamoto S. A Comparison of Techniques for Collecting Skin Microbiome Samples: Swabbing Versus Tape-Stripping. Front Microbiol. 2018 Oct 2;9:2362. doi: 10.3389/fmicb.2018.02362. eCollection 2018. PMID 30333815
- [Result] Lee HJ, Jeong SE, Lee S, Kim S, Han H, Jeon CO. Effects of cosmetics on the skin microbiome of facial cheeks with different hydration levels. Microbiologyopen. 2018 Apr;7(2):e00557. doi: 10.1002/mbo3.557. Epub 2017 Nov 29. PMID 29193830